CLINICAL TRIAL: NCT03812588
Title: Developing New Clinical Management Strategies for Antidepressant Treatments
Brief Title: Contact: Developing New Clinical Management Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor in Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7738
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Clinical Frequency Management: Placebo (Placebo Comparator): Study visits monthly (Week 0, 4, and 8), with phone visits every other week (Week 2 and 6). Double-blind, placebo-controlled treatment with escitalopram 10mg/day, raised to 20mg/day, if non-responders at week 4. If they respond, will be treated in a 3-month Continuation Phase with monthly site visits.
  Interventions: Drug: Placebo
- Research Frequency Management: Placebo (Placebo Comparator): Weekly study visits, treatment with double-blind, placebo controlled escitalopram 10 mg/day, raised to 20mg/day at week 4 if non-responders. If they respond, will be treated in a 3-month Continuation Phase with monthly site visits.
  Interventions: Drug: Placebo
- Clinical Frequency Management: Escitalopram (Active Comparator): Study visits monthly (Week 0, 4, and 8), with phone visits every other week (Week 2 and 6). Double-blind, placebo-controlled treatment with escitalopram 10mg/day, raised to 20mg/day, if non-responders at week 4. If they respond, will be treated in a 3-month Continuation Phase with monthly site visits.
  Interventions: Drug: Escitalopram
- Research Frequency Management: Escitalopram (Active Comparator): Weekly study visits, treatment with double-blind, placebo controlled escitalopram 10 mg/day, raised to 20mg/day at week 4 if non-responders. If they respond, will be treated in a 3-month Continuation Phase with monthly site visits.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram is a Selective Serotonin Reuptake Inhibitor (SSRI) medication that appears to help with symptoms of depression by increasing the availability of specific chemicals in the brain.
  Other Names: Lexapro
  Arms: Clinical Frequency Management: Escitalopram; Research Frequency Management: Escitalopram
Drug: Placebo — A placebo (or dummy pill) is an inert (inactive) substance, typically a tablet, capsule or other dose form that does not contain an active drug ingredient.
  Arms: Clinical Frequency Management: Placebo; Research Frequency Management: Placebo

SUMMARY:
The goal of this study is to develop new methods of administering antidepressant medications that will result in improved drug/placebo separation in randomized controlled trials (RCTs) for Major Depressive Disorder (MDD) and enhanced medication response in open clinical treatment. The highly intensive, weekly visit schedule followed in most antidepressant RCTs radically differs from how antidepressant medications are prescribed in standard clinical practice and is believed to be a major reason why the majority of studies submitted to the Food and Drug Administration (FDA) fail to show a significant difference between medication and placebo. Moreover, a "one size fits all" approach to psychopharmacologic management (i.e., weekly visits for all patients) does not take into account differences between patients that may predispose some individuals to respond positively to frequent follow-up visits, while others may respond negatively or not at all. Clinic visits comprise multiple components that may be therapeutic for depression, including activating patients' behavior, exposing them to medical procedures, permitting social interactions with research staff, and providing supportive meetings with clinicians. Two independent meta-analyses have associated more frequent study visits with increased antidepressant and placebo response as well as decreased separation between medication and placebo. Despite the high costs and potential disadvantages of weekly follow-up visits for patients receiving antidepressant medication, this clinical management strategy has not been studied prospectively to date. It is unknown whether weekly follow-up visits are needed to ensure treatment compliance and patient safety in clinical trials and to what degree contacts with clinicians influence medication and placebo response.

DETAILED DESCRIPTION:
This study utilizes a 2 x 2, double-blind, acute, prospective design randomizing adult

outpatients with MDD to "Research Frequency Management" (RFM, weekly study visits) vs. "Community Frequency Management" (CFM, every 4 weeks study visits) and antidepressant medication vs. placebo. Specifying visit frequency as the independent variable in this study has the distinct advantages of being easily operationalized for research purposes avoiding a priori assumptions about which components of study visits influence antidepressant and placebo response (i.e., behavioral activation vs. doctor-patient relationship vs. medical procedures). Close monitoring of all subjects will be assured by telephone evaluations of individuals randomized to CFM at intervals between monthly visits, and additional study contacts will be scheduled as necessary to maintain patient safety (all extra-protocol contacts will be recorded and included as a variable in outcome analyses). Additionally, subjects will be characterized extensively on clinical, demographic, and psychological measures to pilot the study assessment battery and search for predictor variables influencing the effects of contact frequency on medication and placebo response.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria Method of Ascertainment

1. Men and women aged 18-75 years 1. Clinical interview
2. Diagnosis with Diagnostic and Statistical Manual (DSM) V Major Depressive Disorder (MDD) 2. Clinical interview, Structured Clinical Interview for DSM-V
3. 24-item Hamilton Rating Scale for Depression (HRSD) score ≥ 16 and ≤ 28; 17-item Hamilton Rating Scale for Depression (HRSD) score < 25 3. HRSD by trained rater
4. Capable of providing informed consent and complying with study procedures 4. Clinical interview
5. Using appropriate contraceptive method if woman of child-bearing age and not currently pregnant 5. Clinical interview

Exclusion Criteria:

1. Current comorbid Axis I DSM V disorder other than Mild Substance Use Disorder, Adjustment Disorder, Anxiety Disorder or Personality Disorder 1. Clinical interview, SCID
2. Diagnosis of Moderate to Severe Substance Use Disorder within the past 12 months 2. Clinical interview, SCID, Urine tox
3. present or past history of psychosis, psychotic disorder, mania, or bipolar disorder 3. Clinical interview, SCID
4. baseline HRSD 24-item score > 28 or HRSD suicide item > 2 or baseline HRSD 17-item score ≥ 25 4. HRSD by trained rater
5. History of allergic or adverse reaction to escitalopram, or non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20mg) during the current episode 5. Clinical interview
6. Current treatment with psychotherapy, antidepressants, antipsychotics, or mood stabilizers 6. Clinical interview
7. CGI-Severity score of 6 or greater at baseline 7. CGI based on Clinical interview
8. Acute, severe, or unstable medical illness 8. Clinical interview, Physical Exam, Screening Labs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 29 subjects were enrolled. Of the 29 enrolled, 4 subjects did not continue in the study after enrolling. These 4 subjects did not appear for their randomization visit at which they would have been assigned to a study arm. Thus, 29 patients enrolled and 25 patients started.
Period: Overall Study
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram
Started | 5 | 7 | 5 | 8
Completed | 3 | 5 | 3 | 8
Not Completed | 2 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram | Total
Number analyzed (Participants) | 5 | 7 | 5 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 1
  Between 18 and 65 years | 4 | 5 | 0 | 5 | 14
  >=65 years | 1 | 2 | 4 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (14.40) | 58 (7.26) | 58.8 (22.95) | 60 (13.77) | 58.32 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 4 | 15
  Male | 1 | 3 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 7 | 4 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 3 | 9
  White | 2 | 3 | 3 | 4 | 12
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 7 | 5 | 8 | 25
Hamilton Rating Scale for Depression [Mean (Standard Deviation); unit: units on a scale] — Scale for depressive symptoms administered by trained rater. The Hamilton is the standard measure of depression severity for clinical trials of antidepressants and was chosen to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. The scoring is based on the first 24 items of the Hamilton.
  Sum of the scores of the first 24 items (range from 0 to 74):
  0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
  units on a scale | 18 (4.53) | 20.4 (2.07) | 19.6 (3.65) | 20.8 (4.43) | 19.88 (3.68)
Hamilton Anxiety Rating Scale 14-item Scale [Mean (Standard Deviation); unit: units on a scale] — Scale for anxiety symptoms administered by trained rater. The Hamilton Anxiety is a standard measure of anxiety severity in pharmacotherapy studies that has been shown to have acceptable reliability and validity in studies of depressed patients. Each of the 14 items is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
  units on a scale | 10.2 (3.27) | 9.57 (2.15) | 11.4 (4.22) | 9.62 (2.83) | 10.08 (2.96)
Clinical Global Impressions Severity [Mean (Standard Deviation); unit: units on a scale] — Scales developed to measure the clinician's view of subjects' global functioning before and after initiating a study medication. The Clinical Global Impressions correlates well with other standard outcome measures for depression (e.g., HRSD), is sensitive to change in antidepressant trials, and offers clinically understandable anchor points.
  7-point scale: 0 = Not assessed,
  1 = Normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately ill, 5 = Markedly ill, 6 = Severely ill, 7 = Among the most extremely ill patients
  units on a scale | 4 (0.71) | 4 (0) | 4 (0) | 4 (0.54) | 4 (0.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hamilton Rating Scale for Depression 24-Item Scale to Study Completion (8 Weeks)
Description: Scale for depressive symptoms administered by trained rater. The Hamilton is the standard measure of depression severity for clinical trials of antidepressants and was chosen as the primary outcome measure over other depression rating scales to ensure compatibility of study results with our meta-analyses and ongoing studies of expectancy. The scoring is based on the first 24 items of the Hamilton.
  Sum of the scores of the first 24 items (range from 0 to 74):
  0-7 = NORMAL 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression >=23 = Very Severe Depression
Time Frame: Up to 8 Weeks
Population: Two CFM, Placebo, two RFM, Placebo, and two CFM, Escitalopram participants did not complete the Hamilton Rating Scale for Depression at Week 8, and so their change from baseline Hamilton Rating scale for Depression score could not be calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram
Number analyzed (Participants) | 3 | 5 | 3 | 8
score on a scale | 1.33 (3.51) | 11.4 (4.04) | 5.33 (13.65) | 9.25 (9.21)
Statistical Analysis 1: Comparison: Clinical Frequency Management: Placebo vs Research Frequency Management: Placebo vs Clinical Frequency Management: Escitalopram vs Research Frequency Management: Escitalopram; Test type: Superiority; p = 0.292, Regression, Linear — Linear regression model of condition in predicting change in HRSD-24. P-value and coefficient are Medication:Track. Medication (Escitalopram or Placebo) with Track (RFM or CFM) as co-variates. The threshold for statistical significance was p>0.05; Slope = 7.900, Standard Error of Mean 7.261

2. Secondary Outcome: Change From Baseline Hamilton Anxiety Rating Scale 14-item Scale
Description: Scale for anxiety symptoms administered by trained rater. The Hamilton Anxiety is a standard measure of anxiety severity in pharmacotherapy studies that has been shown to have acceptable reliability and validity in studies of depressed patients. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Up to 8 Weeks
Population: Two CFM, Placebo, two RFM, Placebo, and three CFM, Escitalopram participants did not complete the Hamilton Anxiety at Week 8, and so their change from baseline Hamilton Anxiety score could not be calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram
Number analyzed (Participants) | 3 | 5 | 2 | 8
score on a scale | 3.67 (2.52) | 4.40 (4.22) | 6.50 (4.95) | 3.37 (4.98)

3. Other Pre Specified Outcome: Change From Baseline Clinical Global Impressions
Description: Scales developed to measure the clinician's view of subjects' global functioning before and after initiating a study medication. The Clinical Global Impressions correlates well with other standard outcome measures for depression (e.g., HRSD), is sensitive to change in antidepressant trials, and offers clinically understandable anchor points.
  7-point scale: 0 = Not assessed 4 = Moderately ill
  1 = Normal, not at all ill 5 = Markedly ill 2 = Borderline mentally ill 6 = Severely ill 3 = Mildly ill 7 = Among the most extremely ill patients
Time Frame: Up to 8 Weeks
Population: Two CFM, Placebo, two RFM, Placebo, and two CFM, Escitalopram participants did not complete the CGI at Week 8, and so their change from baseline CGI score could not be calculated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram
Number analyzed (Participants) | 3 | 5 | 3 | 8
score on a scale | 1.00 (1.73) | 1.20 (0.84) | 0.67 (1.15) | 1.50 (1.31)

ADVERSE EVENTS:
Time Frame: Subjects were monitored over a period of 8 weeks.
Description: Subjects in the CFM group were evaluated by study personnel no less frequently than every 2 weeks for 8 weeks. Subjects were monitored for adverse effects, and dose adjustments will be made if indicated during this period of time.
Arm/Group | Clinical Frequency Management: Placebo | Research Frequency Management: Placebo | Clinical Frequency Management: Escitalopram | Research Frequency Management: Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/5 | 1/8
Other Adverse Events (participants affected / at risk) | 2/5 | 6/7 | 1/5 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Frequency Management: Placebo (N=5) | Research Frequency Management: Placebo (N=7) | Clinical Frequency Management: Escitalopram (N=5) | Research Frequency Management: Escitalopram (N=8)
Dehydration (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Frequency Management: Placebo (N=5) | Research Frequency Management: Placebo (N=7) | Clinical Frequency Management: Escitalopram (N=5) | Research Frequency Management: Escitalopram (N=8)
Anorexia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diaphoresis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (15)
Dizziness (General disorders) | 1 (1) | 0 (0) | 1 (6) | 1 (1)
Drowsiness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Excitement (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Headache (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Memory Loss (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orgasm Delay (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Frequency/Urgency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vivid Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight Gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to challenges associated with the pandemic, the study was completed with a smaller sample size than originally intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03812588/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT03812588/SAP_001.pdf